CLINICAL TRIAL: NCT03281369
Title: A Phase Ib/II, Open-Label, Multicenter, Randomized, Umbrella Study Evaluating the Efficacy and Safety of Multiple Immunotherapy-Based Treatment Combinations in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Cancer or Esophageal Cancer (Morpheus-Gastric and Esophageal Cancer)
Brief Title: A Study of Multiple Immunotherapy-Based Treatment Combinations in Patients With Locally Advanced Unresectable or Metastatic Gastric or Gastroesophageal Junction Cancer (G/GEJ) or Esophageal Cancer (Morpheus-Gastric and Esophageal Cancer)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Halozyme Therapeutics (Industry); BioLineRx, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YO39609; 2016-004529-17 (EudraCT Number)
Record Dates: First submitted 2017-09-11; First posted 2017-09-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Gastric Adenocarcinoma or Gastroesophageal Junction Adenocarcinoma or Esophageal Carcinoma
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Fluorouracil; Leucovorin; Oxaliplatin; atezolizumab; cobimetinib; Ramucirumab; Paclitaxel; PEGPH20; 4-fluorobenzoyl-TN-14003; Linagliptin; Cisplatin; Tiragolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- 1L-Control: mFOLFOX6 (Gastric Cancer) (Active Comparator): Participants in the 1L Gastric Cancer Control arm will receive modified FOLFOX6 (mFOLFOX6) treatment consisting of 5-fluorouracil (5-FU), leucovorin (folinic acid), and oxaliplatin. Participants who progressed on treatment may have the option of receiving Atezolizumab + Cobimetinib treatment, provided they meet the eligibility criteria. No longer enrolling participants as of June 2018.
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Oxaliplatin
- 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer) (Experimental): Participants in the 1L-A Gastric Cancer arm will receive mFOLFOX6 treatment consisting of 5-FU, leucovorin and oxaliplatin in combination with atezolizumab plus cobimetinib. No longer enrolling participants as of June 2018.
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Oxaliplatin; Drug: Atezolizumab; Drug: Cobimetinib
- 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer) (Experimental): Participants in the 1L-A2 Gastric Cancer arm will receive mFOLFOX6 treatment consisting of 5-FU, leucovorin and oxaliplatin in combination with atezolizumab during cycles 1 and 2 followed by atezolizumab plus cobimetinib during cycles 3 and beyond. No longer enrolling participants as of June 2018.
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Leucovorin; Drug: Oxaliplatin; Drug: Atezolizumab; Drug: Cobimetinib
- 2L-Control: Ramucirumab + Paclitaxel (Gastric Cancer) (Active Comparator): Participants in the 2L Gastric Cancer Control arm received ramucirumab plus paclitaxel. Participants who progressed on treatment had the option of receiving Atezolizumab + Cobimetinib treatment, provided they met the eligibility criteria. Enrollment completed as of October 2019.
  Interventions: Biological: Ramucirumab; Drug: Paclitaxel
- 2L-1: Atezo + Cobi (Gastric Cancer) (Experimental): Participants in the 2L-1 Gastric Cancer arm received atezolizumab in combination with cobimetinib. Enrollment completed as of October 2019.
  Interventions: Drug: Atezolizumab; Drug: Cobimetinib
- 2L-2: Atezo + PEGPH20 (Gastric Cancer) (Experimental): Participants in the 2L-2 Gastric Cancer arm received atezolizumab in combination with PEGylated recombinant human hyaluronidase (PEGPH20). Participants who progressed on treatment had the option of receiving Atezolizumab + Cobimetinib treatment, provided they met the eligibility criteria. Enrollment completed as of October 2019.
  Interventions: Biological: PEGylated recombinant human hyaluronidase (PEGPH20); Drug: Atezolizumab
- 2L-3: Atezo + BL-8040 (Gastric Cancer) (Experimental): Participants in the 2L-3 Gastric Cancer arm received atezolizumab in combination with BL-8040. Participants who progressed on treatment had the option of receiving Atezolizumab + Cobimetinib treatment, provided they met the eligibility criteria. Enrollment completed as of October 2019.
  Interventions: Drug: BL-8040; Drug: Atezolizumab
- 2L-4: Atezo + Linagliptin (Gastric Cancer) (Experimental): Participants in the 2L-4 Gastric Cancer arm received atezolizumab in combination with linagliptin. Participants who progressed on treatment had the option of receiving Atezolizumab + Cobimetinib treatment, provided they met the eligibility criteria. Enrollment completed as of October 2019.
  Interventions: Drug: Linagliptin; Drug: Atezolizumab
- 1L-1:Atezo+Tiragolumab+Cisplatin+5FU(Esophageal Cancer Cohort) (Experimental): Participants in the 1L-1 Esophageal Cancer arm will receive atezolizumab in combination with tiragolumab and chemotherapy.
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: Tiragolumab; Drug: 5-Fluorouracil (5-FU)
- 1L-2: Atezo+Cisplatin+5-FU (Esophageal Cancer Cohort) (Experimental): Participants in the 1L-2 Esophageal Cancer arm will receive atezolizumab in combination with chemotherapy.
  Interventions: Drug: Atezolizumab; Drug: Cisplatin; Drug: 5-Fluorouracil (5-FU)
- 1L-Control: Cisplatin+5-FU (Esophageal Cancer Cohort) (Active Comparator): Participants in the 1L-Control Eophageal Cancer arm will receive chemotherapy.
  Interventions: Drug: Cisplatin; Drug: 5-Fluorouracil (5-FU)
- 1L-3: Atezo+Tiragolumab (Esophageal Cancer Cohort) (Experimental): Participants in the 1L-3 Esophageal Cancer arm will receive atezolizumab + tiragolumab treatment. Participants from the cisplatin + 5-FU esophageal cancer cohort arm may be permitted to enroll in this arm if they progress after receiving chemotherapy.
  Interventions: Drug: Atezolizumab; Drug: Tiragolumab

INTERVENTIONS:
Drug: 5-Fluorouracil (5-FU) — 5-FU 2400 milligrams per square meter (mg/m^2) by continuous intravenous (IV) infusion over 46 hours on Days 1 and 2 and Days 15 and 16 of every 28-day cycle.
  Arms: 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer); 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer); 1L-Control: mFOLFOX6 (Gastric Cancer)
Drug: Leucovorin — Leucovorin: 100 mg/m^2 IV over 2 hours on Days 1 and 15 of every 28-day cycle.
  Other Names: Folinic acid
  Arms: 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer); 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer); 1L-Control: mFOLFOX6 (Gastric Cancer)
Drug: Oxaliplatin — Oxaliplatin: 100 mg/m^2 administered by IV infusion over 2 hours on Days 1 and 15 of every 28-day cycle.
  Arms: 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer); 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer); 1L-Control: mFOLFOX6 (Gastric Cancer)
Drug: Atezolizumab — Atezolizumab: 840 mg by IV infusion on Days 1 and 15 of every 28-day cycle.
  Other Names: Tecentriq
  Arms: 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer); 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer); 2L-1: Atezo + Cobi (Gastric Cancer)
Drug: Cobimetinib — Cobimetinib: 60 mg by mouth once a day on Days 1-21 of every 28-day cycle
  Other Names: Cotellic
  Arms: 1L-A2: Atezo+mFOLFOX6 followed by Atezo+Cobi (Gastric Cancer); 2L-1: Atezo + Cobi (Gastric Cancer)
Biological: Ramucirumab — Ramucirumab: 8 mg/kg administered by IV infusion over 60 minutes on Days 1 and 15 of every 28-day cycle.
  Arms: 2L-Control: Ramucirumab + Paclitaxel (Gastric Cancer)
Drug: Paclitaxel — Paclitaxel: 80 mg/m^2 administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
  Arms: 2L-Control: Ramucirumab + Paclitaxel (Gastric Cancer)
Biological: PEGylated recombinant human hyaluronidase (PEGPH20) — PEGPH20: 3 micrograms per kilogram (mcg/kg) administered by IV infusion on Days 1, 8, and 15 of every 21-day cycle.
  Arms: 2L-2: Atezo + PEGPH20 (Gastric Cancer)
Drug: BL-8040 — BL-8040: 1.25 mg/kg administered by subcutaneous (SC) injection on Days 1-5 during the 5-day priming period prior to Cycle 1; 1.25 mg/kg administered by SC injection three times a week (Days 1, 3, 5, 8, 10, 12, 15, 17, and 19 of every 21-day cycle).
  Arms: 2L-3: Atezo + BL-8040 (Gastric Cancer)
Drug: Linagliptin — Linagliptin: 5 mg orally once a day of every 21-day cycle.
  Arms: 2L-4: Atezo + Linagliptin (Gastric Cancer)
Drug: Atezolizumab — Atezolizumab: 1200 mg administered by IV infusion on Day 1 of every 21-day cycle
  Other Names: Tecentriq
  Arms: 1L-1:Atezo+Tiragolumab+Cisplatin+5FU(Esophageal Cancer Cohort); 1L-2: Atezo+Cisplatin+5-FU (Esophageal Cancer Cohort); 1L-3: Atezo+Tiragolumab (Esophageal Cancer Cohort); 2L-2: Atezo + PEGPH20 (Gastric Cancer); 2L-3: Atezo + BL-8040 (Gastric Cancer); 2L-4: Atezo + Linagliptin (Gastric Cancer)
Drug: Cobimetinib — Cobimetinib: 40 or 60 mg (depending on the recommended dose determined during the safety run-in phase) by mouth once a day on Days 1-21 of every 28-day cycle.
  Other Names: Cotellic
  Arms: 1L-A: mFOLFOX6 + Atezo + Cobi (Gastric Cancer)
Drug: Cisplatin — Cisplatin: 80 mg/m^2 administered by IV infusion on Day 1 of each 21 day cycle. Treatment will be capped after 6 doses.
  Arms: 1L-1:Atezo+Tiragolumab+Cisplatin+5FU(Esophageal Cancer Cohort); 1L-2: Atezo+Cisplatin+5-FU (Esophageal Cancer Cohort); 1L-Control: Cisplatin+5-FU (Esophageal Cancer Cohort)
Drug: Tiragolumab — Tiragolumab: 600 mg administered by IV infusion on Day 1 of every 21 day cycle.
  Other Names: RO7092284
  Arms: 1L-1:Atezo+Tiragolumab+Cisplatin+5FU(Esophageal Cancer Cohort); 1L-3: Atezo+Tiragolumab (Esophageal Cancer Cohort)
Drug: 5-Fluorouracil (5-FU) — 5-FU 800 mg/m^2 administerd by IV infusion on Days 1-5 of each 21 day cycle.
  Arms: 1L-1:Atezo+Tiragolumab+Cisplatin+5FU(Esophageal Cancer Cohort); 1L-2: Atezo+Cisplatin+5-FU (Esophageal Cancer Cohort); 1L-Control: Cisplatin+5-FU (Esophageal Cancer Cohort)

SUMMARY:
A Phase Ib/II, open label, multi-center, randomized study designed to assess the safety, tolerability, pharmacokinetics and preliminary anti-tumor activity of immunotherapy-based treatment combinations in patients with locally advanced unresectable or metastatic G/GEJ cancer (hereafter referred to as gastric cancer) and esophageal cancer. Two cohorts of patients with gastric cancer have been enrolled in parallel in this study: the second-line (2L) Gastric Cancer Cohort consists of patients with gastric cancer who have progressed after receiving a platinum-containing or fluoropyrimide-containing chemotherapy regimen in the first-line setting, and the first-line (1L) Gastric Cancer Cohort consists of patients with gastric cancer who have not received prior chemotherapy in this setting. In each cohort, eligible patients will be assigned to one of several treatment arms. Additionally, a cohort of patients with esophageal cancer who have not received prior systemic treatment for their disease will be enrolled in this study. Eligible patients will be randomized to chemotherapy or the combination of chemotherapy with checkpoint inhibitor immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

Gastric Cancer Cohorts Inclusion Criteria:

* Age >/= 18 years;
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
* Life expectancy >/= 3 months, as determined by the investigator;
* Histologically or cytologically confirmed locally advanced unresectable or metastatic adenocarcinoma of gastric or gastroesophageal junction; (for the 1L Gastric Cancer Cohort: no prior systemic therapy for the locally advanced or metastatic disease; for the 2L Gastric Cancer Cohort: disease progression during or following a first-line platinum-containing or fluoropyrimidine-containing chemotherapy regimen);
* Availability of a representative tumor specimen that is suitable for determination of PD-L1 and TIGIT levels by IHC and/or additional biomarker status by means of retrospective central testing;
* Only for the 1L Gastric Cancer Cohort: human epidermal growth factor receptor 2 (HER2)-negative tumors;
* Measurable disease (at least one target lesion) according to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1);
* Adequate hematologic and end organ function based on laboratory results obtained within 14 days prior to initiation of study treatment;
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures as outlined for each specific treatment arm;
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as outlined for each specific treatment arm.

Esophageal Cancer Cohort Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of squamous cell carcinoma or adenocarcinoma of the esophagus in locally advanced or metastatic disease;
* No prior systemic treatment for esophageal cancer, with the following exception:

For patients treated with chemotherapy in the locally advanced setting: occurrence of metastasis after 6 months from the last dose of chemotherapy;

* For patients with adenocarcinoma: absence of HER2 expression;
* Life expectancy >/=3 months as determined by the investigator;
* Measurable disease per RECIST v1.1;
* Adequate hematologic and end-organ function;
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating eggs;
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm;
* ECOG Performance Status of 0, 1, or 2.

Exclusion Criteria:

Exclusion criteria for the 2L Gastric Cancer Cohort:

* Urinary protein is > 1 + on dipstick and the required following 24-hour urine collection shows urinary protein > 2000 mg;
* Serious or non-healing wound, peptic ulcer, or bone fracture within 28 days prior to initiation of study treatment;
* History of gastrointestinal perforation and/or fistulae within 6 months prior to initiation of study treatment;
* Presence of a bowel obstruction, history or presence of inflammatory enteropathy, or extensive intestinal resection, Crohn disease, ulcerative colitis, or chronic diarrhea;
* Uncontrolled arterial hypertension >/= 150/ >/= 90 millimeter of mercury (mmHg) despite standard medical management;
* Chronic therapy with non-steroidal anti-inflammatory agents or other anti-platelet agents.

Gastric Cancer Exclusion Criteria:

* Uncontrolled hypercalcemia or symptomatic hypercalcemia requiring continued use of bisphosphonate therapy;
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases;
* History of leptomeningeal disease;
* Active or history of autoimmune disease or immune deficiency;
* History of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan;
* Positive test for human immunodeficiency virus (HIV) at screening;
* Active hepatitis B virus (HBV) or hepatitis C (HCV) infection;
* Severe infection within 4 weeks prior to initiation of study treatment;
* Significant cardiovascular disease;
* Significant bleeding disorder;
* Prior allogeneic stem cell or solid organ transplantation;
* Major surgical procedure, other than for diagnosis, within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the study;
* Treatment with anticoagulation with warfarin, low-molecular-weight heparin, or similar agents for therapeutic purposes;
* History of malignancy other than gastric or gastroesophageal junction carcinoma within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death;
* Known allergy or hypersensitivity to any of the study drugs or their excipients.

Esophageal Cancer Cohort Exclusion Criteria:

* High risk for developing esophageal fistula by clinical assessment or imaging;
* Symptomatic, untreated, or actively progressing central nervous system (CNS) Metastases;
* Positive EBV viral capsid antigen IgM test at screening;
* History of leptomeningeal disease;
* Active or history of autoimmune disease or immune deficiency;
* History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan;
* Active tuberculosis;
* Significant cardiovascular disease within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina;
* History of malignancy other than esophageal cancer within 2 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death;
* Pregnancy or breastfeeding, or intention of becoming pregnant during study treatment or within 5 months after the final dose of atezolizumab or within 90 days after the final dose of tiragolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Objective Response, as Determined by Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) | From Randomization until disease progression or loss of clinical benefit (up to approximately 3-6 years)
Percentage of Participants with Adverse Events (AEs) | From first study treatment administration until 30 days after the last dose or until initiation of new systemic anti-cancer therapy, whichever occurs first (up to approximately 3-6 years)
For Arm 1L-A : Percentage of Participants with Serious and Non-serious Treatment-related AEs | During the safety run-in phase up to 28 days

SECONDARY OUTCOMES:
Progression-Free Survival (PFS), as Determined by Investigator According to RECIST v1.1 | From randomization up to the first occurrence of disease (up to approximately 3-6 years)
Overall Survival (OS) | From randomization up to death from any cause (up to approximately 3-6 years)
Percentage of Participants Who Are Alive at Month 6 and at Month 12 | Month 6, Month 12
Duration of Response, as Determined by Investigator According to RECIST v1.1 | From the date of first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 3-6 years)
Percentage of Participants With Disease Control, as Determined by the Investigator per RECIST v1.1 | From randomization until disease progression or loss of clinical benefit (up to approximately 3-6 years)
Serum Concentration of Atezolizumab | Pre-infusion (0 hour [hr]), 30 minutes (min) post-infusion (infusion=60 min) on Day 1 of Cycle 1; pre-infusion (0 hr) on Day 1 of Cycles 2, 3, 4, 8, 12, 16 (each cycle=28 days); 30 days and 120 days after last dose (up to approximately 3-6 years)
Plasma Concentration of Cobimetinib | Prior to cobimetinib dose, 2-4 hr after cobimetinib dose on Day 15 of Cycle 1 (cycle length=28 days)
Plasma Concentration of PEGPH20 | Pre-infusion (0 hr) on Day 1 of Cycle 1 up to 30 days and 120 days after last dose (up to approximately 3-6 years) (Detailed timeframe is provided in outcome measure description)
  Pre-infusion (0 hr), 5 min and 1-3 hrs post infusion (infusion duration=10-12 min) on Day 1 of Cycle 1; pre-infusion (0 hr) on Days 8 and 15 of Cycle 1, Day 1 of Cycles 3, 4, 8, 12, 16; pre-infusion (0 hr) and 5 min post-infusion on Day 1 of Cycle 2 (each cycle=21 days); 30 days and 120 days after last dose (up to approximately 3-6 years)
Plasma Concentration of BL-8040 | Pre-dose (0 hr) on Day 1 of priming period (1 week prior to Day 1 of Cycle 1) up to 30 days after last dose (up to approximately 3-6 years) (Detailed timeframe is provided in outcome measure description)
  Pre-dose (0 hr) on Day 1 of priming period (1 week prior to Day 1 of Cycle 1); 1 hr post-dose on Days 1, 5 of priming period; pre-dose (0 hr), 1 hour post-dose on Day 15 of Cycle 1 and Day 1 of Cycles 2, 3, 4, 8, 12, 16; pre-dose (0 hr) on Day 1 of Cycle 20 and every 4 cycles thereafter (each cycle=21 days) (up to approximately 3-6 years); 30 days after last dose (up to approximately 3-6 years)
Plasma Concentration of Linagliptin | 2 hr postdose oral linagliptin on Day 1 of Cycle 1, prior to atezolizumab infusion and predose oral linagliptin on Day 15 of Cycle 1 as well as on Day 1 of Cycles 2, 3, and 4
Percentage of Participants With Anti-Drug Antibody (ADA) to Atezolizumab | Pre-infusion (0 hr) on Day 1 of Cycles 1, 2, 3, 4, 8, 12, 16 (each cycle=28 days); 30 days and 120 days after last dose (up to approximately 3-6 years)
Percentage of Participants With ADA to PEGPH20 | Pre-infusion (0 hr) on Day 1 of Cycles 1, 2, 3, 4, 8, 12, 16 (each cycle=21 days); 30 days and 120 days after last dose (up to approximately 3-6 years)
Percentage of Participants With ADA to BL-8040 | Pre-dose (0 hr) on Day 1 of priming period (1 week prior to Day 1 of Cycle 1) up to 30 days after last dose (up to approximately 3-6 years) (Detailed timeframe is provided in outcome measure description)
  Pre-dose (0 hr) on Day 1 of priming period (1 week prior to Cycle 1 Day 1), Day 15 of Cycle 1 and Day 1 of Cycles 2, 3, 4, 8, 12, 16, 20 and every 4 cycles thereafter (each cycle=21 days) (up to approximately 3-6 years); 30 days after last dose (up to approximately 3-6 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (6):
  - Mayo Clinic Cancer Center, Scottsdale, Arizona
  - Uni of Southern California, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Santa Monica, California
  - Columbia University Medical Center, New York, New York
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Blacktown Hospital, Blacktown, New South Wales
  - Monash Medical Centre-Moorabbin Campus, Clayton, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Israel (2):
  - Rambam Health Care Campus, Haifa
  - Sourasky Medical Centre, Tel Aviv
- South Korea (7):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital (SNUH) - Medical Oncology Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University College of Medicine (YUCM)-Yonsei Cancer Center, Seoul
  - University of Ulsan College of Medicine - Asan Medical Center (AMC) - Asan Cancer Center (ACC), Songpa-gu
  - The Catholic University of Korea St. Vincent's Hospital, Suwon
- Spain (2):
  - Universidad de Navarra - Clinica Universitaria de Navarra (CUN), Pamplona, Navarre
  - Hospital Universitari Vall dHebron, Barcelona
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital (NTUH) - Cancer Research Center, Zhongzheng Dist.
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Barts and The London School of Medicine and Dentistry - Barts Cancer Institute (BCI)-CECM, London
  - The Royal Marsden, London
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust - Royal Marsden Hospital (RMH) - Sutton, Sutton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Sun JM, Chao Y, Kim SB, Rha SY, Evans TRJ, Strickland AH, Wainberg Z, Chau I, Pelles-Avraham S, Ajani J, Malhotra R, Liu Q, Li S, Cha E, Kalaitzidou M, Huang X, Allen S, Hsu CH. First-line tiragolumab plus atezolizumab and chemotherapy in patients with previously untreated, locally advanced unresectable or metastatic oesophageal cancer (MORPHEUS-EC): a randomised, open-label, phase 1b/2 trial. Lancet Oncol. 2026 Jan;27(1):90-102. doi: 10.1016/S1470-2045(25)00402-4. PMID 41449151
- [Derived] Ko AH, Kim KP, Siveke JT, Lopez CD, Lacy J, O'Reilly EM, Macarulla T, Manji GA, Lee J, Ajani J, Alsina Maqueda M, Rha SY, Lau J, Al-Sakaff N, Allen S, Lu D, Shemesh CS, Gan X, Cha E, Oh DY. Atezolizumab Plus PEGPH20 Versus Chemotherapy in Advanced Pancreatic Ductal Adenocarcinoma and Gastric Cancer: MORPHEUS Phase Ib/II Umbrella Randomized Study Platform. Oncologist. 2023 Jun 2;28(6):553-e472. doi: 10.1093/oncolo/oyad022. PMID 36940261